CLINICAL TRIAL: NCT05734378
Title: Prognosis of Cerebral Small Vessel Disease - a Prospective Cohort Study (PRO-SVD)
Brief Title: Prognosis of Cerebral Small Vessel Disease
Acronym: PRO-SVD
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02535
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Amyloid Angiopathy; Small Vessel Cerebrovascular Disease; Cadasil; CAA - Cerebral Amyloid Angiopathy
Keywords: small vessel disease; CAA; cerebral amyloid angiopathy; hypertensive arteriopathy; deep perforator arteriopathy; CADASIL
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Cerebral Small Vessel Diseases; CADASIL; Cerebral Amyloid Angiopathy, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prognosis of small vessel disease (SVD) depends on the underlying type of SVD and index manifestation.

The aim of this prospective, observational cohort study is to determine the risk of different outcome events among patients with SVD according to the type of index presentation.

ELIGIBILITY:
Inclusion Criteria:

* Hypertensive deep perforator arteriolopathy (DPA), clinically symptomatic with either ICH, ischaemic stroke, cognitive impairment or severe radiological manifestation (Fazekas ≥II)
* Cerebral amyloid angiopathy (CAA according to modified Boston or Edinburgh criteria), clinically symptomatic with either ICH (including cSAH), amyloid spells, cognitive impairment or severe radiological manifestation (CMB≥2)
* Other SVD (i.e. CADASIL or other sporadic or genetic SVD)

Exclusion Criteria:

* Life expectancy of <6 months due to not-SVD related causes (i.e. cancer)
* Patient is unlikely to attend follow-up visits

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospectively recruited cohort of patients treated with cerebral small vessel disease at Inselspital Bern University Hospital. Patients are recruited at the emergency department, neurology in-patient ward, Stroke Unit, IMC, ICU and outpatient clinics.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
Intracerebral haemorrhage (ICH) | 1 year
  Non-traumatic, intracerebral haemorrhage (ICH, including convexity subarachnoid haemorrhage)
Ischaemic stroke | 1 year
  Defined by CT and/or MRI
Cardio-vascular death | 1 year
  According to the treating physician

SECONDARY OUTCOMES:
Other intracranial bleeding | 1 year
  Subdural haematoma, subarachnoid haemorrhage
Other (transient) neurological attacks | 1 year
  Including transient ischaemic attack (TIA), transient neurological attack (TNA), amyloid spells, (focal) seizures
Cognitive impairment | 1 year
  Montreal Cognitive Assessment (MoCA, range 0-30 points) < 26 points (corresponding to impaired cognitive function) and/or new impairment in activities of daily living as defined by the treating physician.
New-onset of extracranial vascular disease | 1 year
  As judged by the treating physician
Functional outcome | 1 year
  Modified Rankin scale score (ordinal score, range 0-6, a score of 0 corresponds to no symptoms at all, while a score of 6 corresponds to death)

CONTACTS AND LOCATIONS:
Overall Officials: David J Seiffge, Prof, MD, Principal Investigator — Department of Neurology, Inselspital Bern University Hospital
Locations (1):
- Department of Neurology, Inselspital Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided